CLINICAL TRIAL: NCT00623909
Title: Laser Therapy in the Treatment of Post Thoracotomy Pain; A Pilot Study.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left the institution
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0709009417
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Laser Therapy; Post Thoracotomy Pain
Keywords: Laser Therapy; Post Thoracotomy Pain; AvicennaTM laser

STUDY DESIGN:
Masking Description: Not applicable, study terminated prior to enrollment and closed.
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): To demonstrate the safety of the AvicennaTM class IV laser for application over the skin of human subjects. This study was terminated prior to subject enrollment and closed.
  Interventions: Device: AvicennaTM class IV laser application

INTERVENTIONS:
Device: AvicennaTM class IV laser application — AvicennaTM class IV laser for application over the skin of human subjects in the treatment of post-thoracotomy pain syndrome. Six sessions, twenty minutes applications over a period of six weeks.

SUMMARY:
The purpose of this study is to demonstrate the safety of the AvicennaTM class IV laser for application over the skin of human subjects. In addition, we seek to measure the effectiveness and utility of this class 4 laser therapy in the treatment of post-thoracotomy pain syndrome.

DETAILED DESCRIPTION:
This study was terminated prior to enrollment and closed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 25-65 years old with chest wall pain after lung surgery lasting more than 2 months after surgery.
* Subjects shall have failed conservative treatment which may include rest, physical therapy, braces, and over the counter anti-inflammatory medications. All those enrolled will be native English speakers and have at least a high school degree

Exclusion Criteria:

* Subjects will be excluded if they are pregnant (which will be confirmed by a urine pregnancy test if they are of childbearing age)
* Have previous history of other pain syndromes or psychiatric disorders.
* We will exclude the morbidly obese (BMI >30) because the laser may not be able to penetrate deep enough through adipose tissue. In addition, subjects who have had previous back surgery, or are on antidepressants for the treatment of depression in the preceding 6 weeks will be excluded as these may represent potential confounding factors.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The McGill pain questionnaire | 6 Treatments/6 Weeks

SECONDARY OUTCOMES:
The visual analog scale | 6 Weeks
An infrared thermometer will measure skin temperature before and after the treatment | 6 Treatments/6 Weeks
A 4-point Likert scale (none, mild, moderate, and severe) will be used to document skin redness. | 6 Treatments/6 Weeks
A 4-point Likert scale (none, mild, moderate, and severe) will be used to document skin tenderness | 6 Treatments/6 Weeks
At the end of the study patients will rate their satisfaction with the treatment using an 11 point Likert scale where 0 means completely dissatisfied and 10 means completely satisfied. | 6 Treatments/6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edward Rubin, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Not Applicable, study terminated prior to enrollment and closed